CLINICAL TRIAL: NCT00199654
Title: PET Interest in the Follow Up of Colorectal Cancer Stage II and III: Phase III Randomised Study
Brief Title: Positron Emission Tomography (PET) Interest in the Follow Up of Colorectal Cancer Stage II and III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: I03001
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer stage II and III
MeSH Terms: conditions — Colorectal Neoplasms

INTERVENTIONS:
Procedure: PET

SUMMARY:
The follow up of colorectal cancer after curative surgery has to find loco-regional relapses or synchronous metastases, and to detect adenomas and new cancer on the rest of the colon.

The increase of survival after relapse of the colorectal cancer depends on the possibility of curative action or after chemotherapy response.

This is a Phase III open-labeled, multicenter, multidisciplinary, randomised study, comparing 2 arms of 188 patients (i.e. 376 total patients).

Study Period (date of first inclusion/last inclusion): 3 years.

Follow Up: 3 years.

The primary objective is the evaluation of PET performance in the earlier relapse detection of the colorectal cancer relapse in comparison with conventional control (including carcinoembryonic [CEA] levels and other classic radiological exams).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Confirmed stage II or III (TNM)
* Patient with curative surgery for colorectal adenocarcinoma
* Total digestive endoscopy prior or post surgery.
* Age > 18 years old
* Normal liver ultrasound and chest X-ray or thoraco-abdomino pelvic computed tomography (CT) scan.
* In fertile women, efficient contraception or postmenopausal patient (amenorrhea for at least 1 year)

Exclusion Criteria:

* Serious concomitant pathology
* Uncontrolled diabetes with a classical treatment (glycaemia >1.4 g/l)
* Other malignant tumour within the last 5 years (except for curatively treated basocellular carcinoma of the skin or in situ cervical carcinoma).
* Uncontrolled infection
* Women who are pregnant or lactating
* Inability to understand informed consent
* Psychological or geographic impossibility to follow up for three years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2004-02; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Time to colorectal cancer relapse

SECONDARY OUTCOMES:
Evaluation of overall survival in the two groups | after curative resection of colorectal cancer stage II or III
Evaluation of the rate of curative surgery | after relapse
Comparison of the medical cost in the two detection strategies

CONTACTS AND LOCATIONS:
Overall Officials: Nicole TUBIANA-MATHIEU, MD, Principal Investigator — University Hospital, Limoges
Locations (5):
- France (5):
  - Cancérologie et Hépato-Gastro-Entérologie, Bordeaux
  - Institut François Baclesse, Caen
  - Médecine Nucléaire, Limoges
  - Oncologie Médicale, Limoges
  - Oncologie Digestive, Marseille

REFERENCES:
- [Derived] Monteil J, Le Brun-Ly V, Cachin F, Zasadny X, Seitz JF, Mundler O, Selvy M, Smith D, Rullier E, Lavau-Denes S, Lades G, Labrunie A, Lecaille C, Valli N, Leobon S, Terrebonne E, Deluche E, Tubiana-Mathieu N. Comparison of 18FDG-PET/CT and conventional follow-up methods in colorectal cancer: A randomised prospective study. Dig Liver Dis. 2021 Feb;53(2):231-237. doi: 10.1016/j.dld.2020.10.012. Epub 2020 Nov 2. PMID 33153929